CLINICAL TRIAL: NCT01440712
Title: Prospective Randomized Double Blind Study of the Effect of Gastrografin on Postoperative Ileus After Colorectal Surgery
Brief Title: Study of the Effect of Water Soluble Oral Contrast (Gastrografin) on Postoperative Ileus After Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Sebastiano Biondo, Principal investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ileus_gastro; 2010-024096-87 (EudraCT Number)
Record Dates: First submitted 2011-09-21; First posted 2011-09-26 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Ileus
Keywords: Gastrografin; Postoperative ileus; Colo-rectal surgery; Effects on morbidity and mortality of postoperative ileus
MeSH Terms: interventions — Diatrizoate Meglumine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastrografin (Experimental): Patients located in this group will be treated with the administration of 100 ml of gastrografin by the nasogastric tube, only once, after the diagnosis of postoperative ileus.
  Interventions: Drug: Gastrografin
- physiological serum (Placebo Comparator): Patients included in this group will be treated with 100 ml of physiological serum 0,9% by the nasogastric tube, only once, after the diagnosis of postoperative ileus.
  Interventions: Drug: physiological serum

INTERVENTIONS:
Drug: Gastrografin — Administration of 100 ml of gastrografin by the nasogastric tube, only once.
  Arms: Gastrografin
Drug: physiological serum — Administration of 100 ml of physiological serum 0,9% by the nasogastric tube, only once.
  Arms: physiological serum

SUMMARY:
The purpose of this trial is to determine whether the water-soluble contrast (gastrografin) is more effective in the treatment of postoperative ileus than the conventional one.

ELIGIBILITY:
Inclusion Criteria:

* All patients with postoperative ileus after colorectal surgery, defined as the presence from the third postoperative day, abdominal distension, nausea, vomiting with or without abdominal pain or discomfort by dilation of bowel loops, confirmed radiology of the abdomen, and which are: Age > 18 years Patients undergoing laparotomy or laparoscopy for the following variants of colorectal disease with or without stoma:

  1. Neoplasia.
  2. Inflammatory disease.
  3. Diverticular disease. Patients who have been treated with standard PCA as postoperative analgesia. Signed informed consent. Undergoing elective or scheduled

Exclusion Criteria:

* Patient's refusal to sign informed consent
* Pregnancy or lactation
* Hypersensitivity to iodinated contrast agents (it´s the only contraindication to oral Gastrografin) Presence of other problems that justify the etiology of postoperative ileus:

  1. Anastomotic leakages.
  2. Mesenteric vascular disease.
  3. Incarcerated hernias.
  4. Intra-abdominal abscesses or collections.
  5. Metabolic or electrolyte disturbances. If during the course of the study one of the reasons previously cited as the etiology of postoperative ileus is present, the patient shall also be excluded. Also excluded patients undergoing emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to resolution of postoperative ileus after surgery defined as time to tolerance of oral intake of solid or semisolid food | While the patient is admitted to the hospital. An average of 11 days since the intervention.

SECONDARY OUTCOMES:
Hospital stay after diagnosis of ileus | While the patient is admitted to the hospital. An average of 11 days since the intervention.
  Postoperative complications were assessed in the intervening period between the immediate postoperative phase and when the patient is discharged.
Percentage of patients requiring total parenteral nutrition. | While the patient is admitted to the hospital. An average of 11 days since the intervention
  Postoperative complications were assessed in the intervening period between the immediate postoperative phase and when the patient is discharged
Presence of postoperative pain and analgesic required | While the patient is admitted to the hospital. An average of 11 days since the intervention
  Postoperative complications were assessed in the intervening period between the immediate postoperative phase and when the patient is discharged
Percentage of mortality during hospitalization. | While the patient is admitted to the hospital. An average of 11 days since the intervention
  Postoperative complications were assessed in the intervening period between the immediate postoperative phase and when the patient is discharged

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, Dr., Principal Investigator — Bellvitge University Hospital
Locations (3):
- Spain (3):
  - Hospital Universitari de la Vall d´Hebron, Barcelona, Barcelona
  - Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Girona, Girona, Girona

REFERENCES:
- [Background] Chen JH, Hsieh CB, Chao PC, Liu HD, Chen CJ, Liu YC, Yu JC. Effect of water-soluble contrast in colorectal surgery: a prospective randomized trial. World J Gastroenterol. 2005 May 14;11(18):2802-5. doi: 10.3748/wjg.v11.i18.2802. PMID 15884127
- [Background] Biondo S, Pares D, Mora L, Marti Rague J, Kreisler E, Jaurrieta E. Randomized clinical study of Gastrografin administration in patients with adhesive small bowel obstruction. Br J Surg. 2003 May;90(5):542-6. doi: 10.1002/bjs.4150. PMID 12734858
- [Background] Abbas SM, Bissett IP, Parry BR. Meta-analysis of oral water-soluble contrast agent in the management of adhesive small bowel obstruction. Br J Surg. 2007 Apr;94(4):404-11. doi: 10.1002/bjs.5775. PMID 17380561
- [Background] Delaney CP, Wolff BG, Viscusi ER, Senagore AJ, Fort JG, Du W, Techner L, Wallin B. Alvimopan, for postoperative ileus following bowel resection: a pooled analysis of phase III studies. Ann Surg. 2007 Mar;245(3):355-63. doi: 10.1097/01.sla.0000232538.72458.93. PMID 17435541
- [Background] Waldhausen JH, Schirmer BD. The effect of ambulation on recovery from postoperative ileus. Ann Surg. 1990 Dec;212(6):671-7. doi: 10.1097/00000658-199012000-00004. PMID 2256758
- [Background] Bohm B, Milsom JW, Fazio VW. Postoperative intestinal motility following conventional and laparoscopic intestinal surgery. Arch Surg. 1995 Apr;130(4):415-9. doi: 10.1001/archsurg.1995.01430040077017. PMID 7710343
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Derived] Biondo S, Miquel J, Espin-Basany E, Sanchez JL, Golda T, Ferrer-Artola AM, Codina-Cazador A, Frago R, Kreisler E. A Double-Blinded Randomized Clinical Study on the Therapeutic Effect of Gastrografin in Prolonged Postoperative Ileus After Elective Colorectal Surgery. World J Surg. 2016 Jan;40(1):206-14. doi: 10.1007/s00268-015-3260-9. PMID 26446450